CLINICAL TRIAL: NCT06431724
Title: A Prospective Analysis of Adherence to National Cervical Cancer Screening Recommendations in Women Age >65
Brief Title: A Review of Cervical Cancer Screening Practices in Women Age >65
Status: Enrolling by invitation | Type: Observational
Sponsor: Sarasota Memorial Health Care System (Other)
Responsible Party: Principal Investigator, Tamela Fonseca, Director of Research, Sarasota Memorial Health Care System
Other Study IDs: 23-ONC-34
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Cervical Cancer
Keywords: cervical cancer screening; cervical cancer; geriatric cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women >65 years who are considered at risk of developing cervical cancer: 200 women >65 years who are considered at risk of developing cervical cancer.
  Interventions: Other: Patient Survey
- Primary care providers and gynecologic providers: 100 Licensed Primary Care and Gynecologic Providers which includes APRNs, PAs, and Physicians.
  Interventions: Other: Provider Survey

INTERVENTIONS:
Other: Patient Survey — A simple data intake collection from the patients regarding their medical history that will allow the researchers to assess if recommended guidelines were followed.
  Groups: Women >65 years who are considered at risk of developing cervical cancer
Other: Provider Survey — A survey will be used to evaluate providers' practices, knowledge and adherence to guidelines, and decision making related to current practice for cervical screening in women >65.
  Groups: Primary care providers and gynecologic providers

SUMMARY:
The goal of this research study is to examine adherence to national guidelines for cervical cancer screening in women age >65. Patient surveys will provide information about women age >65 current cervical screening practices and allow researchers to compare that information to national recommended guidelines regarding cervical screenings. Provider surveys will provide information from surveyed providers about screening knowledge and current provider practices for women patients > 65 for cervical cancer. The results may be used to make future recommendations for improving gynecological care and to help develop effective strategies for ensuring guideline adherence.

DETAILED DESCRIPTION:
This prospective study will be conducted to determine adherence to the national guidelines for cervical cancer screening in women >65. A nonpaired patient and provider survey will be utilized to assess both provider and patient adherence to the national cervical cancer screening guidelines. Providers who meet study eligibility will be asked to complete a survey containing questions regarding their current practice for cervical cancer screening, the guidelines they follow, and their decision-making process when deciding who to screen. Patients who meet study eligibility will be asked to complete a survey detailing the frequency and types of cervical cancer screenings they have had and any relevant outcomes. The aims of the study are to assess cervical cancer screening practices among at risk women age >65 years and describe adherence to nationally recommended cervical cancer screening guidelines for this same patient group and among primary care providers (PCPs) and gynecologists. To assess adherence, the Sarasota Memorial Research Institute (SMRI) will conduct a research study which includes patients age >65 from the Sarasota Memorial Health Care System (SMHCS) and their First Physician's Group (FPG) affiliates and providers. Patients who agree to participle will be surveyed to determine their behaviors surrounding cervical cancer screenings. Primary care physicians and gynecologists who are either members of the American Academy of Family Physicians (AAFP), ACOG, or practice within SMHCS or FPG providers who agree to participate will also receive a separate one-time survey to assess adherence to the ACOG, ACS, and USPSTF guidelines for conducting cervical cancer screenings. The target survey sample size for this study will be 200 patients, women >65 years who are considered at risk of developing cervical cancer (women with a history of a hysterectomy will be excluded) and receive gynecological services at SMHCS. In addition, 100 primary care physicians (PCPs) and gynecologists will be targeted.

ELIGIBILITY:
For participants:

Inclusion Criteria:

* Women age >65 who have not had a hysterectomy.
* Women who received gynecological services within the SMHCS/FPG network FPG physician offices -Primary Care or Gynecologic Care))

Exclusion Criteria:

* Woman has a history of prior hysterectomy.
* Woman is age 65 years and under
* Woman does not receive gynecologic services within SMHCS/FPG network.

For providers:

Inclusion Criteria:

* Licensed Primary Care and Gynecologic Providers which includes APRNs, PAs, and Physicians.
* Provider practices in the U.S.
* Provider performs gynecological screenings as part of their current practice.

Exclusion Criteria:

* Provider does not practice in the United States.
* Provider does not provide gynecological screenings.
* Provider does not have an active license as a Primary Care Provider or Gynecologic Provider (APRNs, PAs, or Physicians).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sample size for this study will consist of 200 patients and 100 providers who are comprised of PCPs and gynecologists affiliated with the American Academy of Family Physicians (AAFP) or the American College of Obstetricians and Gynecologists (ACOG) or who are practitioners within SMHCS/FPG locations.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-07-28 (Estimated); Study Completion 2024-07-28 (Estimated)

PRIMARY OUTCOMES:
Exact binomial 95% confidence intervals will be used. | Both patient and provider surveys are one-time only events. Their participation is limited to only the single time they take the survey which is estimated to take approximately 15 minutes.
  To report adherence to national guidelines within each group, exact binomial 95% confidence intervals will be used. A multi-variant analysis will be conducted to determine the frequency, types, and outcomes of cervical cancer screening/s performed and patient and provider characteristics associated with guideline adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Tamela Fonseca, PhD, RN, CCRC, Principal Investigator — Sarasota Memorial Health Care System Research Institute
Locations (1):
- Sarasota Memorial Health Care System, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arbyn M, Weiderpass E, Bruni L, de Sanjose S, Saraiya M, Ferlay J, Bray F. Estimates of incidence and mortality of cervical cancer in 2018: a worldwide analysis. Lancet Glob Health. 2020 Feb;8(2):e191-e203. doi: 10.1016/S2214-109X(19)30482-6. Epub 2019 Dec 4. PMID 31812369
- [Background] Bujang MA, Omar ED, Baharum NA. A Review on Sample Size Determination for Cronbach's Alpha Test: A Simple Guide for Researchers. Malays J Med Sci. 2018 Nov;25(6):85-99. doi: 10.21315/mjms2018.25.6.9. Epub 2018 Dec 28. PMID 30914882
- [Background] Dilley S, Huh W, Blechter B, Rositch AF. It's time to re-evaluate cervical Cancer screening after age 65. Gynecol Oncol. 2021 Jul;162(1):200-202. doi: 10.1016/j.ygyno.2021.04.027. Epub 2021 Apr 26. PMID 33926748
- [Background] Feldman S, Cook E, Davis M, Gershman ST, Hanchate A, Haas JS, Perkins RB. Cervical Cancer Incidence Among Elderly Women in Massachusetts Compared With Younger Women. J Low Genit Tract Dis. 2018 Oct;22(4):314-317. doi: 10.1097/LGT.0000000000000435. PMID 30256336
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Mills JM, Morgan JR, Dhaliwal A, Perkins RB. Eligibility for cervical cancer screening exit: Comparison of a national and safety net cohort. Gynecol Oncol. 2021 Aug;162(2):308-314. doi: 10.1016/j.ygyno.2021.05.035. Epub 2021 Jun 3. PMID 34090706
- [Background] Qin J, Shahangian S, Saraiya M, Holt H, Gagnon M, Sawaya GF. Trends in the use of cervical cancer screening tests in a large medical claims database, United States, 2013-2019. Gynecol Oncol. 2021 Nov;163(2):378-384. doi: 10.1016/j.ygyno.2021.08.023. Epub 2021 Sep 8. PMID 34507826
- [Background] Saslow D, Solomon D, Lawson HW, Killackey M, Kulasingam SL, Cain J, Garcia FA, Moriarty AT, Waxman AG, Wilbur DC, Wentzensen N, Downs LS Jr, Spitzer M, Moscicki AB, Franco EL, Stoler MH, Schiffman M, Castle PE, Myers ER; American Cancer Society; American Society for Colposcopy and Cervical Pathology; American Society for Clinical Pathology. American Cancer Society, American Society for Colposcopy and Cervical Pathology, and American Society for Clinical Pathology screening guidelines for the prevention and early detection of cervical cancer. Am J Clin Pathol. 2012 Apr;137(4):516-42. doi: 10.1309/AJCPTGD94EVRSJCG. PMID 22431528
- [Background] Surveillance, Epidemiology, and End Results (SEER) Cancer Stat Facts: Cervix uteri Cancer, n.d.
- [Background] Tsang S, Royse CF, Terkawi AS. Guidelines for developing, translating, and validating a questionnaire in perioperative and pain medicine. Saudi J Anaesth. 2017 May;11(Suppl 1):S80-S89. doi: 10.4103/sja.SJA_203_17. PMID 28616007
- [Background] Yost S, Hoekstra A. Cervical cancer in women over 65: An analysis of screening. Gynecol Oncol Rep. 2018 May 22;25:48-51. doi: 10.1016/j.gore.2018.05.010. eCollection 2018 Aug. PMID 30023421
- See also: ACOG Updated Cervical Cancer Screening Guidelines — https://www.acog.org/clinical/clinical-guidance/practice-advisory/articles/2021/04/updated-cervical-cancer-screening-guidelines
- See also: U.S. Census Bureau (2022). QuickFacts — http://www.census.gov/quickfacts/sarasotacountyflorida.
- See also: United States Preventative Task Force (USPTF). Cervical Cancer Screening. August 21, 2018. — http://www.uspreventiveservicestaskforce.org/uspstf/recommendation/cervical-cancer-screening